CLINICAL TRIAL: NCT02139397
Title: A Phase I/II Trial of DFMO in Combination With Bortezomib in Patients With Relapsed or Refractory Neuroblastoma
Brief Title: Study of Difluoromethylornithine (DFMO) in Combination With Bortezomib for Relapsed or Refractory Neuroblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: Beat NB Cancer Foundation (Other); Because of Ezra (Other); K C Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMTRC010
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Results first posted 2024-04-25 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma Recurrent
MeSH Terms: interventions — Eflornithine; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DFMO and Bortezomib (Experimental): Subjects will take DFMO by mouth 2 times a day for each day of a 21 day cycle and Bortezomib will be given by IV push on days 1, 4, and 8 of each 21 day cycle.
  Interventions: Drug: DFMO; Drug: Bortezomib

INTERVENTIONS:
Drug: DFMO
  Other Names: D,L-ɑdifluoromethylornithine; Eflornithine
Drug: Bortezomib
  Other Names: Velcade

SUMMARY:
The purpose of this research study is to evaluate an investigational drug (DFMO) in combination with bortezomib, for relapsed and refractory neuroblastoma. DFMO is an investigational drug because it has not been approved by the U.S. Food and Drug Administration (FDA). This study will look at the safety and tolerability of DFMO in combination with bortezomib as well as the tumors response to this study drug.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≤ 21 years at the time of diagnosis.
* Diagnosis: Histologic verification at either the time of original diagnosis or relapse of neuroblastoma.
* Disease Status: For the purposes of this study, aggressive multidrug chemotherapy is defined as chemotherapy including 2 or more agents that must include an alkylating agent and a platinum-containing compound. Patients must have one of the following:
* First episode of recurrent disease following completion of aggressive multi-drug frontline therapy.
* First episode of progressive disease during aggressive multi-drug frontline therapy.
* Primary resistant/refractory disease detected at the conclusion of at least 4 cycles of aggressive multidrug induction chemotherapy on or according to a high-risk neuroblastoma protocol (examples include Children's Oncology Group trials: A3973, ANBL0532, ANBL09P1, etc.).
* Measurable or evaluable disease, including at least one of the following: Measureable tumor by CT or MRI; or A positive meta-iodobenzylguanidine (MIBG) or positron emission computed tomography (PET) scan; or Positive bone marrow biopsy/aspirate.
* Current disease state must be one for which there is currently no known curative therapy or no additional therapies proven to prolong survival with an acceptable quality of life.
* A negative urine pregnancy test is required for female subjects of child bearing potential (onset of menses or ≥13 years of age).
* Organ Function Requirements:

  1. Subjects must have adequate liver function as defined by:

     * AST (aspartate aminotransferase) and alanine aminotransferase (ALT) <5x upper limit of normal
     * Serum bilirubin must be ≤ 2.0 mg/dl
  2. Subjects must have adequate Bone Marrow function defined as:

For patients without bone marrow involvement:

* Peripheral absolute neutrophil count (ANC) ≤ 750/uL
* Platelet count 50,000/uL (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment. Exception: Patients that are platelet dependent due to previous extensive treatment- e.g. - MIBG therapy).
* Hemoglobin ≥ 8.0 g/dL (may receive red blood cell transfusions) Patients known to have bone marrow involvement with neuroblastoma are eligible provided that minimum ANC and platelet count criteria are met but are not evaluable for hematological toxicity.

  * Subjects must have adequate renal function defined as: Serum creatinine based on age/gender.
  * Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* Lansky score <50%
* BSA (body surface area) body surface body surface m2 of <0.25
* Prior Therapy- Patients must have fully recovered from the acute toxic effects of all prior anti- cancer chemotherapy and be within the following timelines:

  1. Myelosuppressive chemotherapy: Must not have received within 2 weeks of enrollment onto this study (6 weeks if prior nitrosourea).
  2. Hematopoietic growth factors: At least 5 days since the completion of therapy with a growth factor.
  3. Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the Study Chair.
  4. Immunotherapy: At least 6 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines.
  5. Monoclonal antibodies: At least 7 days or 3 half-lives, whichever is longer, must have elapsed since prior treatment with a monoclonal antibody.
  6. Radiotherapy: At least 14 days since the last treatment except for radiation delivered with palliative intent to a non-target site.
  7. Stem Cell Transplant or Rescue: No evidence of active graft vs. host disease and ≥ 2 months must have elapsed since transplant.
* Investigational Drugs: Subjects who have received another investigational drug within the last 14 days are excluded from participation.
* Infection: Subjects who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Neville, MD, Study Chair — Children's Mercy Hospital Kansas City
Locations (6):
- United States (6):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children- MD Anderson, Orlando, Florida
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- See also: Beat Childhood Cancer Consortium website — http://www.beatcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Difluoromethylornithine (DFMO) 1500 mg/m^2; Phase I: DFMO 2000 mg/m^2; Phase I: DFMO 2500 mg/m^2: Subjects will take DFMO by mouth 2 times a day for each day of a 21 day cycle and Bortezomib will be given by IV push on days 1, 4, and 8 of each 21 day cycle.
- Phase 2: The highest tolerated DFMO dose from the Phase I dose escalation will be used for the Phase II portion of the study. Subjects will receive oral DFMO twice daily on each day of this 21-day cycle along with Bortezomib and Etoposide.
Period: Overall Study
Arm/Group | Phase I: Difluoromethylornithine (DFMO) 1500 mg/m^2 | Phase I: DFMO 2000 mg/m^2 | Phase I: DFMO 2500 mg/m^2 | Phase 2
Started | 3 | 7 | 6 | 0
Completed | 3 | 7 | 6 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that took at least one dose of study drug
Groups:
- Phase I: DFMO 1500 mg/m^2; Phase I: DFMO 2000 mg/m^2"; Phase I: DFMO 2500 mg/m^2": Subjects will take DFMO by mouth 2 times a day for each day of a 21 day cycle and Bortezomib will be given by IV push on days 1, 4, and 8 of each 21 day cycle.
- Total: Total of all reporting groups
Arm/Group | Phase I: DFMO 1500 mg/m^2 | Phase I: DFMO 2000 mg/m^2" | Phase I: DFMO 2500 mg/m^2" | Phase 2 | Total
Number analyzed (Participants) | 3 | 7 | 6 | 0 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 7 | 6 | 0 | 16
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 10 [8 to 11] | 7.1 [3 to 14] | 10 [6 to 18] |  | 8.75 [3 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 |  | 5
  Male | 2 | 5 | 4 |  | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 |  | 2
  Not Hispanic or Latino | 2 | 7 | 4 |  | 13
  Unknown or Not Reported | 0 | 0 | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0
  Asian | 0 | 0 | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 0 | 1 |  | 1
  White | 3 | 7 | 3 |  | 13
  More than one race | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Phase I- To determine the safety and tolerability of DFMO in combination with bortezomib at 3 dose levels of DFMO: 1500mg/m2 twice daily, 2000mg/m2 twice daily, and 2500mg/m2 twice daily in subjects with relapsed or refractory neuroblastoma who receive one full cycle of this dose.
  Phase II- Study did not enroll to Phase II. Study completed at end of Phase I.
Time Frame: Adverse Events were collected starting with the date of the first dose of study drug until 30 days after last dose of study drug, ongoing related adverse events were continued to be followed until resolution, on average 6 months.
Population: All subjects that took at least one dose of DFMO
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: DFMO 1500 mg/m^2 | Phase I: DFMO 2000 mg/m^2" | Phase I: DFMO 2500 mg/m^2" | Phase 2
Number analyzed (Participants) | 3 | 7 | 6 | 0
Participants | 2 | 1 | 3 |

2. Secondary Outcome: Determine the Overall Response Rate (ORR) of Participants Using RECIST Criteria
Description: To determine the overall response rate (ORR) by the presence of radiologically assessable disease by cross-sectional imaging and in MIBG (meta-iodobenzylguanidine) or PET (positron emission computed tomography) scans. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI imaging and/or by MIBG or PET scans: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), At least a 20% increase in the sum of the disease measurements for measurable lesions, Stable Disease, Neither sufficient decrease to qualify for PR or sufficient increase to qualify for PD from study entry. Overall Response (OR) = CR + PR.
Time Frame: Followed until off therapy, generally 1 year
Population: Analyzed population only includes evaluable subjects, defined as subjects that made it to an evaluation time point (disease evaluation scans), or had a documented progression of disease prior to evaluation time point.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: DFMO 1500 mg/m^2: Subjects that received Dose level 1 - 1500 mg/m2 BID (twice a day)
- Phase I: DFMO 2000 mg/m^2: Subjects that received Dose level 2 - 2000 mg/m2 BID
- Phase I: DFMO 2500 mg/m^2: Subjects that received Dose level 3 - 2500 mg/m2 BID
- Phase 2: Did not enroll
Arm/Group | Phase I: DFMO 1500 mg/m^2 | Phase I: DFMO 2000 mg/m^2 | Phase I: DFMO 2500 mg/m^2 | Phase 2
Number analyzed (Participants) | 3 | 5 | 5 | 0
Participants
  Complete Response | 0 | 0 | 0 |
  Partial Response | 1 | 0 | 0 |
  Stable Disease | 1 | 2 | 2 |
  Progressive Disease | 1 | 2 | 3 |
  Mixed Response | 0 | 1 | 0 |

3. Secondary Outcome: Determine the Progression Free Survival (PFS) of Participants Using Days Until Progression
Description: Time to progression (PFS), defined as the period from the start of the treatment until the criteria for progression are met taking as reference the screening measurements. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of the disease measurements for measurable lesions, taking as reference the smallest disease measurement recorded since the start of treatment (nadir), and minimum 5 mm increase over the nadir or the appearance of one or more new lesions or appearance of positive bone marrow.
Time Frame: From date of start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Groups:
- Phase I: DFMO 1500 mg/m^2: Subjects that received Dose level 1 - 1500 mg/m2 BID
Arm/Group | Phase I: DFMO 1500 mg/m^2 | Phase I: DFMO 2000 mg/m^2 | Phase I: DFMO 2500 mg/m^2 | Phase 2
Number analyzed (Participants) | 3 | 6 | 5 | 0
Days | 108.3 [41 to 160] | 51.2 [23 to 84] | 61.8 [21 to 140] |

ADVERSE EVENTS:
Time Frame: Adverse Events were collected starting with the date of the first dose of study drug until 30 days after last dose of study drug, ongoing related adverse events were continued to be followed until resolution, on average of 1 year.
Arm/Group | Phase I: DFMO 1500 mg/m^2 | Phase I: DFMO 2000 mg/m^2 | Phase I: DFMO 2500 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/7 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/7 | 1/6
Other Adverse Events (participants affected / at risk) | 2/3 | 1/7 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: DFMO 1500 mg/m^2 (N=3) | Phase I: DFMO 2000 mg/m^2 (N=7) | Phase I: DFMO 2500 mg/m^2 (N=6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: DFMO 1500 mg/m^2 (N=3) | Phase I: DFMO 2000 mg/m^2 (N=7) | Phase I: DFMO 2500 mg/m^2 (N=6)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-04-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT02139397/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT02139397/ICF_001.pdf